CLINICAL TRIAL: NCT05978804
Title: Remote Home-based Electrical Stimulation (tDCS) in Primary Progressive Aphasia (With Frontotemporal Dementia or Alzheimer's Pathology) and Mild Cognitive Impairment/Alzheimer's.
Brief Title: Home-based tDCS in Frontotemporal Dementia or Alzheimer's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Ybrain Inc. (Industry); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NA_00071337-4; R01DC014475 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-08-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Primary Progressive Aphasia; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Aphasia, Primary Progressive; Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects meeting eligibility criteria will be randomized to receive either tDCS + cognitive training or only tDCS. After 50 treatment sessions (approximately 10 weeks) participants will switch to the other condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS on the DLPFC + Cognitive Intervention(s) (Experimental): Participants will receive active tDCS on DLPFC + Cognitive Intervention(s) first and then receive only active tDCS Intervention after a three-month washout period.
  Interventions: Other: Computerized Cognitive Training; Device: Active tDCS (tDCS) on DLPFC
- Active tDCS on the DLPFC only (Experimental): Participants will receive active tDCS on the DLPFC-only intervention first and then receive active tDCS + Cognitive Intervention(s) after a three-month washout period.
  Interventions: Device: Active tDCS (tDCS) on DLPFC

INTERVENTIONS:
Other: Computerized Cognitive Training — Computerized Cognitive training (BrainHQ or Constant Therapy)
  Arms: Active tDCS on the DLPFC + Cognitive Intervention(s)
Device: Active tDCS (tDCS) on DLPFC — Device: Active tDCS on DLPFC Stimulation will be delivered by a constant current stimulator (Mind STIM). The electrical current will be administered to a pre-specified region of the brain (DLPFC). The stimulation will be delivered at an intensity of 2 milliamperes (mA) (estimated current density 0.04 mA/cm2; estimated total charge 0.048 Coulombs/cm2) in a ramp-like fashion for a maximum of 20 minutes.

SUMMARY:
The primary objective of this research is to evaluate the effects of non-invasive brain stimulation and computerized cognitive training on executive functioning in individuals with Primary Progressive Aphasia (PPA), mild cognitive impairment (MCI), or dementia. In this study, investigators will use transcranial direct current stimulation (tDCS) to stimulate the left dorsolateral prefrontal cortex (DLPFC). Previous studies have demonstrated that tDCS over the DLPFC led to improvements in attention deficit caused by stroke, Parkinson's Disease, and major depression as well as language deficits caused by neurodegenerative conditions such as primary progressive aphasia or mild cognitive impairment. The investigators seek to expand on this literature by investigating how anodal tDCS paired with and without cognitive training will impact executive functioning in PPA with Frontotemporal Dementia or Alzheimer's Disease pathology and Mild Cognitive Impairment/Alzheimer's Disease (e.g. shifting, updating, monitoring, and manipulation).

DETAILED DESCRIPTION:
In this within-subject cross-over protocol, all participants will receive both, cognitive training and brain stimulation tDCS. Participants will be randomly assigned to begin with either cognitive training and brain stimulation (dual therapy) or just brain stimulation (monotherapy) and will receive the complementary therapy program in the second round of treatment. During each period of therapy, participants will receive 50 treatment sessions over the course of approximately 10 weeks. The computerized cognitive training and brain stimulation will both be preprogrammed to be done at home by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Must be clinically diagnosed with PPA, fronto-temporal dementia (FTD), MCI or mild Alzheimer's disease (AD). Diagnosis will be based on neuropsychological testing, language testing (most commonly the Western Aphasia Battery), MRI, and clinical assessment.
* Must be right-handed.
* Must be proficient in English.
* Must have a minimum high-school education.

Exclusion Criteria:

* Uncorrected visual or hearing impairment by self-report.
* Stroke/other premorbid neurological disorder affecting the brain.
* Any other developmental language-based learning disorder other than PPA.
* Inability to follow directions for baseline tasks.
* Pre-existing psychiatric disorders such as behavioral disturbances, severe depression, and schizophrenia that do not allow them to comply or follow the study schedule and requirements such as repeated evaluation and therapy will be excluded.

Exclusion Criteria for MRI participation:

* Severe claustrophobia.
* Cardiac pacemakers or ferromagnetic implants.
* Pregnant women.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in language composite outcome | Before intervention, immediately after intervention
  A single language composite outcome will be generated by computing the mean of the z-scores the following oral and written naming, spelling, and sentence comprehension and repetition tasks: Philadelphia Naming Test (Short Form), Boston Naming Test, Hopkins Action Naming Assessment, Hopkins Dysgraphia Battery, National Alzheimer's Coordinating Center Sentence Repetition. The investigators will take the z-score for each task and aggregate them in order to get a composite z-score.
Change in Executive Composite Outcome | Before intervention, immediately after intervention
  A single executive composite will be generated by computing the mean of the z-scores of the tasks below reflecting new learning and memory, processing speed and executive functioning, attention and working memory, and verbal fluency respectively: Rey Auditory Verbal Learning Test, Trail Making Test A and B, Attention Network Task, Digit and Spatial Span, and Category fluency and Verbal Fluency. The investigators will take the z-score for each task and aggregate them in order to get a composite z-score.
Change in Global Cognitive Scores | Before intervention, immediately after intervention
  This will be measured using the Montreal Cognitive Assessment (MoCA). Scored out of 30 points, higher is better.

SECONDARY OUTCOMES:
Change in Selective attention and cognitive flexibility | Before intervention, immediately after intervention
  This will be measured using the Attention Network Task (ANT). An efficiency score for executive attention is derived by comparing scores on trials with congruent flankers to trials with incongruent flankers. Subjects will tend to be slower and less accurate for incongruent trials, the size of the different indicates the extent to which an individual can supress conflicting response tendencies. A larger difference between congruent and incongruent trials score indicates a lower executive efficiency.
Change in attention and task switching | Before intervention, immediately after intervention
  This will be measured using Trail Making Task and N-Back (2-back) scores. The Trail Making Test is scored by time. Less time needed to complete the task is indicative of better task-switching. The N-back task is a well-established task that assesses working memory and working memory capacity. Participants are presented with words in sequence and instructed to reply whether the current word matches the one presented 2 words ago. Scoring will be based on the total number of correct responses (hit rate) minus the number of incorrect responses (false alarm rate), where a greater score is better.
Change in working memory capacity. | Before intervention, immediately after intervention
  This will be measured using Digit Span Backward for verbal working memory and spatial span Backward for spatial working memory. The digit span backward is a well-established task that assesses rote immediate verbal memory and working memory. Participants are presented with a series of digits and are instructed to repeat the digits in the reverse order. The spatial span task is an analog to the Digit Span Task, but instead the participants are presented with an array of squares which are sequentially presented and must be touched in the same order. For both tasks scoring is based on the number of digits or blocks shown in a trial (i.e. 1,7 is 2 digits). There are two trials for each span, if both trials are correct the score is a whole number (i.e. 2). If one trial is incorrect in a span, subtract 0.5 from that tier (i.e. 1.5). Increase in score from before to after intervention is considered a benefit.
Change in level of Depressive Symptoms | Before intervention, immediately after intervention
  Measured by the Hamilton Depression Rating Scale (HAM-D) which is a 17-item measure that was designed to assess frequency and intensity of depressive symptoms in patients with Major Depressive Disorder (MDD). This measure contains somatic and suicidal ideation items and has demonstrated reliability, validity, and efficiency in adult populations. Scoring is out of 53, a score of 0-7 is accepted to be normal, a score of 20 or higher indicates at least moderate severity.

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States